CLINICAL TRIAL: NCT02384681
Title: Effects of Auditory Fatigue in Medical Regulation Assistants Working With Headset: Objective Measures
Brief Title: Evaluation of Auditory Fatigue in Medical Regulation Assistants
Acronym: EchoSam
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other); Institut National de Recherche et de Sécurité, Nancy, France (Unknown)
Responsible Party: Principal Investigator, Cecile PARIETTI-WINKLER, University Professor - Hospital Practitioner, Central Hospital, Nancy, France
Other Study IDs: 2014-A01904-43
Record Dates: First submitted 2015-03-05; First posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Auditory Fatigue
Keywords: Speech intelligibility; Short-term memory; Working memory; Perceived mental task load
MeSH Terms: conditions — Speech Intelligibility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exposed: Medical regulation assistants working with headset
  Interventions: Other: Exposure to auditory fatigue
- Non-Exposed: Participants working without headset

INTERVENTIONS:
Other: Exposure to auditory fatigue — 12-hour auditory exposure
  Groups: Exposed

SUMMARY:
Auditory monitoring of employees is currently based on pure-tone audiometry. However, this clinical examination does not prevent from deafness but established it a posteriori. From a preventive standpoint, it is important to detect hearing professional pain before the development of irreversible(s) clinical(s) symptom(s). The investigators' hypothesis is that auditory fatigue results from damages of primary and secondary central auditory pathways involving cognitive processes.

The assessment of auditory fatigue includes the evaluation of speech intelligibility, short-term memory, working memory and perceived mental task load. The main objective of this study is to identify, among regulating medical assistants working with headset, a central auditory fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Participants without hearing loss and without ontological antecedents in the past 5 years
* Participants gave their written informed consent
* Participants are affiliated to the french social welfare
* Preliminary clinical examination

Exclusion Criteria:

* Ontological antecedents in the past 5 years
* Pathology of the external or middle ear
* Abnormality in audiometric examination
* Participants already enrolled in an other research protocol
* Participants covered by articles L.1121-5 à L.1121-8 et L.1122-1-2 of the French Public Health Code

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical regulation assistants working with or without headset
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-10 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change in speech intelligibility | Before and after the 12-hour auditory exposure

SECONDARY OUTCOMES:
Change in perceived mental task load | During (after 2-hour auditory exposure) and after the 12-hour auditory exposure
Change in short-term memory | Before and after the 12-hour auditory exposure
Change in working memory | Before and after the 12-hour auditory exposure

CONTACTS AND LOCATIONS:
Overall Officials: Parietti-Winkler Cécile, MD, PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- University Hospital of Nancy, Nancy, France